CLINICAL TRIAL: NCT04703413
Title: User Satisfaction When Catheterizing With Hydrophilic Urinary Catheters From a More Sustainable Manufacturing Process. An Open, Prospective, Post-market Clinical Follow-up Investigation.
Brief Title: User Satisfaction When Catheterizing With Hydrophilic Urinary Catheters From a More Sustainable Manufacturing Process.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LOF-0036
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Bladder Voiding Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LoFric® OrigoTM or LoFric® SenseTM (Experimental): Hydrophilic male (LoFric Origo) and female (LoFric Sense) urinary catheters for single use. Target subject population are subjects suffering from bladder voiding dysfunction and are experienced in intermittent catheterization (IC).
  Interventions: Device: LoFric® OrigoTM and LoFric® SenseTM

INTERVENTIONS:
Device: LoFric® OrigoTM and LoFric® SenseTM — The investigational device is either a CE-marked LoFric® OrigoTM , 40 cm, CH12/CH14 or LoFric® SenseTM, 15 cm, CH12. They are all intermittent urinary catheters with a Nelaton tip from a more sustainable manufacturing process. All subjects will use the investigational device for 30 days each.

SUMMARY:
An open, prospective, single arm, multicenter clinical investigation. All subjects will use the investigational device for 30 days each.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, subjects must fulfil all of the following criteria:

1. Provision of informed consent i.e. subject must be able to understand and sign the Informed Consent Form
2. Aged 18 years and over, both gender
3. Bladder dysfunction, all diagnosis practicing IC at least 2 times daily
4. Using catheters in the sizes available in the investigation (15 cm, CH 12 or 40 cm CH 12/14, Nelaton tip)
5. Experienced users of IC defined as a minimum of 4 weeks on therapy prior investigation start
6. Adults able to read, write and understand information given to them regarding the investigation

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Ongoing, symptomatic UTI at enrolment as judged by investigator. The definition of UTI, is a positive urine culture of ≥103 CFU/ml of ≥1 bacterial species and presence of symptoms or signs compatible with UTI with no other identified source of infection.
2. Known urethral stricture which, in the opinion of the investigator, could influence the subject's evaluation of the catheters.
3. Involvement in the planning and conduct of the investigation (applies to both Wellspect/site staff).
4. Previous enrolment in the present investigation.
5. Simultaneous participation in another clinical investigation that may impact the primary endpoint.
6. Expected or severe non-compliance to the CIP as judged by the investigator and/or Wellspect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Subjects' satisfaction, when practicing IC (insertion/withdrawal) using study device. | 30 days
  The subject's assessment of satisfaction using a five-level scale in a pPRO (Wellspect Follow-up questionnaire): How satisfied have you been with the catheterization (insertion/withdrawal) when using the investigational device?
  1. = completely unsatisfied
  2. = unsatisfied
  3. = neutral
  4. = satisfied
  5. = completely satisfied

SECONDARY OUTCOMES:
Reason for dissatisfaction (if any) when practicing IC with study device. | 30 days
  The proportion of subjects that are unsatisfied/completely unsatisfied and specifying the reason in free text. pPRO (Wellspect questionnaire)
Experience of any problems before, during and after catheterization with investigational device. | 30 days
  The proportion of subjects that experienced any problems. A yes/no scale, if yes, a specification (free text) is required.
  pPRO (Wellspect questionnaire)
Catheter usability (incl. ease of use) when practicing IC with investigational device. | 30 days
  The mean of all subject's answers/domain score of ISC-Q (ease of use) completed at the end of investigation visits. pPRO (Wellspect questionnaire) and ISC-Q - domain ease of use.
QoL when practicing IC with investigational device. | 30 days
  ISC-Q total mean score The mean of all subjects' total score of ISC-Q completed at the end of investigation visits.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Wittebo, M.Sc. Pharm., Study Director — Wellspect HealthCare; Ruth Kirschner-Hermanns, Univ.-Prof. Dr. med., Principal Investigator — Universitätsklinikum Bonn, Germany; Antje Foresti, Dr. med., Principal Investigator — Zentrum für Kontinenz und Neuro-Urologie, Kliniken Maria Hilf GmbH, Mönchengladbach; Alexander Höinghaus, Dr. med., Principal Investigator — Gemeinschaftspraxis für Urologie, Dierdorf
Locations (3):
- Germany (3):
  - Leitung der Neuro-Urologie Klinik der Urologie und Kinderurologie Universitätsklinikum Bonn, Bonn
  - Gemeinschaftspraxis für Urologie, Dierdorf
  - Zentrum für Kontinenz und Neuro-Urologie Kliniken Maria Hilf GmbH Akademisches Lehrkrankenhaus der Uniklinik RWTH Aachen, Mönchengladbach, Mönchengladbach